CLINICAL TRIAL: NCT01459913
Title: A Phase 3b Study of 2 Treatment Durations of Telaprevir, Peg-IFN (Pegasys®), and Ribavirin (Copegus®) in Treatment-Naive and Prior Relapser Subjects With Genotype 1 Chronic Hepatitis C and IL28B CC Genotype
Brief Title: Efficacy of a 12-Week Regimen of Telaprevir, Pegylated Interferon, and Ribavirin in Treatment-Naive and Prior Relapser Subjects With Interleukin28B (IL28B) CC Genotype
Acronym: CONCISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor on 13 January 2014 due to a decision to modify the drug development plan.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX11-950-114
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis C, Chronic
Keywords: VX-950; INCIVEK; INCIVO
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) (Experimental): Telaprevir 1125 milligram (mg) tablet twice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 12 weeks. Only subjects who completed initial 12 week of telaprevir and Peg-IFN/RBV and met rapid viral response (RVR, undetectable Hepatitis C Virus [HCV] Ribonucleic Acid [RNA] at Week 4) criteria, were randomized in this group, as planned, and did not receive any further treatment.
  Interventions: Drug: Telaprevir; Drug: Pegylated Interferon Alfa-2a; Drug: Ribavirin
- Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) (Experimental): Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 weeks. Only subjects who completed initial 12 week of telaprevir and Peg-IFN/RBV and met RVR criteria, were randomized in this group, as planned.
  Interventions: Drug: Telaprevir; Drug: Pegylated Interferon Alfa-2a; Drug: Ribavirin
- Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) (Experimental): Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 weeks. Only subjects with RVR who permanently discontinued telaprevir, Peg-IFN-alfa-2a, or RBV treatment before Week 12, and had extended rapid viral response (eRVR, undetectable HCV RNA at Weeks 4 and 12), were included in this group, as planned.
  Interventions: Drug: Telaprevir; Drug: Pegylated Interferon Alfa-2a; Drug: Ribavirin
- Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized) (Experimental): Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks. Only subjects with no RVR or no RVR assessment, and subjects with RVR who permanently discontinued telaprevir, Peg-IFN-alfa-2a, or RBV treatment before Week 12, who did not have eRVR or eRVR assessment, were included in this group, as planned.
  Interventions: Drug: Telaprevir; Drug: Pegylated Interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Tablet
  Other Names: INCIVEK; INCIVO; VX-950
Drug: Pegylated Interferon Alfa-2a — Subcutaneous Injection
  Other Names: Pegasys; Peg-IFN-Alfa-2a
Drug: Ribavirin — Tablet
  Other Names: Copegus; RBV

SUMMARY:
The purpose of this study is to evaluate if a 12-week total regimen of telaprevir in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) and ribavirin (RBV) (T12/PR12) is safe and effective in subjects who have the interleukin-28B (IL28B) CC genotype. The subjects enrolled in this study will have chronic hepatitis C virus (HCV) infection and will not have cirrhosis of the liver.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 70 years of age, inclusive
* Treatment-naive OR subjects (prior relapsers) may be included who did not achieve sustained viral response 24 weeks after last planned dose of study drug (SVR24) after at least 1 prior course of Peg-IFN/RBV therapy of standard duration and had a documented undetectable HCV RNA level at the planned end of treatment of at least 42-week duration
* Subjects have IL28B CC genotype determined during screening
* Subjects have genotype 1 chronic hepatitis C and laboratory evidence of HCV infection for at least 6 months, defined by (1) documented HCV serology test at least 6 months before the first screening visit demonstrating the presence of anti-HCV antibody, or (2) documented presence of HCV RNA by a sensitive and specific assay at least 6 months before the first screening visit, or (3) documented histologic evidence of chronic hepatitis C demonstrated by fibrosis on a standardized histologic grading system at least 6 months before the first screening visit. If only inflammation is present in the liver histologic report, then 6 months of laboratory evidence is required

Exclusion Criteria:

* Subjects have received previous treatment with telaprevir or any other protease inhibitor(s) for chronic hepatitis C
* Subjects who did not achieve SVR24 after at least 1 prior course of Peg-IFN/RBV therapy of standard duration and never achieved undetectable HCV RNA while on treatment
* Subjects have evidence of hepatic decompensation
* Subjects have evidence of cirrhosis
* Subjects have diagnosed or suspected hepatocellular carcinoma
* Subjects have any other cause of significant liver disease in addition to hepatitis C, which may include but is not limited to malignancy with hepatic involvement, hepatitis B, drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis, or primary biliary cirrhosis. Steatosis is allowed if clinically asymptomatic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Friedman, M.D., Study Director — Vertex Pharmaceuticals Incorporated
Locations (70):
- United States (46):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - La Jolla, California
  - Los Angeles, California
  - California, Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - California, San Francisco, California
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Bradenton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Baltimore, Maryland
  - Columbia, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Novi, Michigan
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Egg Harbor, New Jersey
  - Vineland, New Jersey
  - Flushing, New York
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Pennsylvania, Hershey, Pennsylvania
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Virginia, Fairfax, Virginia
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Austria (2):
  - Linz
  - Vienna
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
- Germany (8):
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Hanover
  - Leipzig
  - Munich
- Israel (5):
  - Haifa
  - Israel, Jerusalem
  - Nazareth
  - Petah Tikva
  - Tel Litwinsky
- Poland (4):
  - Bialystok
  - Czeladź
  - Mysłowice
  - Wroclaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received telaprevir in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a)/ ribavirin (RBV). Planned duration of telaprevir treatment was 12 weeks. Minimum planned duration of Peg-IFN-alfa-2a/RBV treatment was 12 weeks; however, was dependent on virologic response during initial 12 weeks of telaprevir plus Peg-IFN-alfa-2a/RBV.
Period: Overall Study
Arm/Group | Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized)
Started | 106 | 52 | 19 | 62
Completed | 65 | 32 | 6 | 29
Not Completed | 41 | 20 | 13 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 5
Not completed — Lost to Follow-up | 7 | 4 | 1 | 8
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Non- Compliance | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 30 | 15 | 9 | 11
Not completed — Other | 0 | 0 | 3 | 1
Not completed — Did Not Meet Inclusion Criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis (FA) Set included all subjects who received at least 1 dose of study drug and fulfilled all relevant inclusion criteria. One subject from "Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized)" was excluded from the FA Set due to having HCV Genotype 6.
Groups:
- Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized): Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 12 weeks. Only subjects who completed initial 12 week of telaprevir and Peg-IFN/RBV and met RVR criteria, were randomized in this group, as planned, and did not receive any further treatment.
- Total: Total of all reporting groups
Arm/Group | Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized) | Total
Number analyzed (Participants) | 106 | 52 | 19 | 61 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.82) | 44.8 (12.89) | 54.4 (8.70) | 49.8 (10.56) | 47.4 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 16 | 11 | 29 | 95
  Male | 67 | 36 | 8 | 32 | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sustained Viral Response 12 Weeks After Last Planned Dose of Study Drug (SVR12)
Description: SVR12 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at 12 weeks after last planned dose of study drug. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL) and the lower limit of detection was 10 IU/mL. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: 12 weeks after last planned dose of study drug (up to Week 36)
Population: Full Analysis (FA) Set.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
percentage of participants | 88.7 | 96.2

2. Secondary Outcome: Percentage of Subjects With Sustained Viral Response 4 Weeks After Last Planned Dose of Study Drug (SVR4)
Description: SVR4 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at 4 weeks after last planned dose of study treatment. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL) and the lower limit of detection was 10 IU/mL. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: 4 weeks after last planned dose of study drug (up to Week 28)
Population: FA Set.
Measure: Number; unit: percentage of participants
Groups:
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized): Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 12 weeks. Only subjects who completed initial 12 week of telaprevir and Peg-IFN/RBV and met RVR criteria, were randomized in this group, as planned, and did not receive any further treatment.
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
percentage of participants | 89.6 | 98.1

3. Secondary Outcome: Percentage of Subjects With Sustained Viral Response 24 Weeks After Last Planned Dose of Study Drug (SVR24)
Description: SVR24 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at 24 weeks after last planned dose of study treatment. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL) and the lower limit of detection was 10 IU/mL. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: 24 weeks after last planned dose of study drug (up to Week 48)
Population: FA Set.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
percentage of participants | 85.8 | 92.3

4. Secondary Outcome: Percentage of Subjects With Sustained Viral Response at Week 72 (SVR72)
Description: SVR72 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at Week 72. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL) and the lower limit of detection was 10 IU/mL. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: Week 72
Population: FA Set. Here number of subjects analyzed = subjects who were evaluable for this measure. Subjects who did not have the SVR72 assessment because they discontinued the study due to 'Study Terminated by the Sponsor' are excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 76 | 37
percentage of participants | 72.4 | 86.5

5. Secondary Outcome: Percentage of Subjects With Viral Relapse
Description: Viral relapse was defined as having detectable HCV RNA during antiviral follow-up in subjects who had HCV RNA less than (<) lower limit of quantification (LLOQ) at end of treatment. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The LLOQ was 25 IU/mL and the lower limit of detection was 10 IU/mL. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: After last dose of study drug up to 4 weeks (up to Week 28), 12 weeks (up to Week 36), 24 weeks (up to Week 48) antiviral follow-up
Population: FA Set.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
percentage of participants
  4 Weeks | 1.9 | 0.0
  12 Weeks | 7.5 | 0.0
  24 Weeks | 10.4 | 0.0

6. Secondary Outcome: Percentage of Subjects With On-Treatment Virologic Failure
Description: On-treatment virologic failure was defined as subjects who met futility (as per investigator discretion) or who completed the assigned treatment duration and had detectable HCV RNA at planned end of treatment (up to 48 weeks). This outcome was planned to be assessed in all reporting groups and results were to be reported for total arm as well.
Time Frame: Baseline up to Week 48
Population: FA Set.
Measure: Number; unit: percentage of participants
Groups:
- Telaprevir+Peg-IFN-alfa-2a, RBV (Total): All subjects who received telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, up to 48 weeks.
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized) | Telaprevir+Peg-IFN-alfa-2a, RBV (Total)
Number analyzed (Participants) | 106 | 52 | 19 | 61 | 238
percentage of participants | 0 | 0 | 0 | 3.3 | 0.8

7. Secondary Outcome: Number of Subjects With Rapid Viral Response (RVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. RVR was defined as undetectable HCV RNA 4 weeks after the start of study treatment. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: Week 4
Population: FA Set.
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
participants | 106 | 52

8. Secondary Outcome: Number of Subjects With Extended Rapid Viral Response (eRVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. eRVR was defined as undetectable HCV RNA at both 4 weeks and 12 weeks after the start of study treatment. This outcome was planned to be assessed only in "Telaprevir 12 Week (Wk)+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized)" and "Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)" reporting groups.
Time Frame: Week 4 and Week 12
Population: FA Set.
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized)
Number analyzed (Participants) | 106 | 52
participants | 105 | 51

9. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents administered during the course of the study.
Time Frame: Baseline up to Week 48
Population: Safety set included all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized)
Number analyzed (Participants) | 106 | 52 | 19 | 62
participants
  AEs | 104 | 51 | 19 | 61
  SAEs | 5 | 4 | 3 | 13

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized)
Serious Adverse Events (participants affected / at risk) | 5/106 | 4/52 | 3/19 | 13/62
Other Adverse Events (participants affected / at risk) | 104/106 | 51/52 | 19/19 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) (N=106) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) (N=52) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) (N=19) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized) (N=62)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 7
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abscess oral (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Wk (Randomized) (N=106) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Randomized) (N=52) | Telaprevir 12 Wk+Peg-IFN-alfa-2a,RBV 24 Wk (Non Randomized) (N=19) | Telaprevir 12 Wk +Peg-IFN-alfa-2a,RBV 48 Wk (Non Randomized) (N=62)
Fatigue (General disorders) | 55 | 25 | 12 | 26
Pyrexia (General disorders) | 26 | 13 | 4 | 15
Influenza like illness (General disorders) | 28 | 10 | 8 | 9
Asthenia (General disorders) | 14 | 8 | 3 | 13
Irritability (General disorders) | 9 | 7 | 2 | 9
Chills (General disorders) | 6 | 6 | 0 | 9
Injection site erythema (General disorders) | 5 | 4 | 0 | 3
Pain (General disorders) | 5 | 3 | 1 | 3
Malaise (General disorders) | 0 | 1 | 1 | 5
Oedema peripheral (General disorders) | 1 | 4 | 1 | 1
Chest pain (General disorders) | 2 | 2 | 1 | 0
Injection site reaction (General disorders) | 1 | 1 | 0 | 4
Injection site rash (General disorders) | 1 | 2 | 0 | 2
Chest discomfort (General disorders) | 0 | 4 | 0 | 0
Injection site pruritus (General disorders) | 1 | 2 | 1 | 0
Local swelling (General disorders) | 1 | 1 | 0 | 1
Thirst (General disorders) | 1 | 0 | 1 | 1
Feeling abnormal (General disorders) | 1 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 1
Enanthema (General disorders) | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 49 | 19 | 13 | 33
Diarrhoea (Gastrointestinal disorders) | 19 | 6 | 6 | 11
Vomiting (Gastrointestinal disorders) | 17 | 6 | 6 | 11
Anorectal discomfort (Gastrointestinal disorders) | 22 | 9 | 3 | 5
Anal pruritus (Gastrointestinal disorders) | 10 | 8 | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 8 | 4 | 1 | 6
Dry mouth (Gastrointestinal disorders) | 5 | 3 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 9 | 2 | 1 | 3
Proctalgia (Gastrointestinal disorders) | 5 | 4 | 0 | 3
Constipation (Gastrointestinal disorders) | 4 | 1 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 44 | 17 | 8 | 24
Rash (Skin and subcutaneous tissue disorders) | 31 | 15 | 9 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 11 | 4 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 11 | 6 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2 | 3 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 5 | 1 | 4 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 30 | 16 | 5 | 17
Dizziness (Nervous system disorders) | 17 | 6 | 6 | 14
Dysgeusia (Nervous system disorders) | 13 | 2 | 2 | 5
Hypoaesthesia (Nervous system disorders) | 2 | 5 | 0 | 1
Migraine (Nervous system disorders) | 2 | 3 | 1 | 1
Disturbance in attention (Nervous system disorders) | 3 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 3 | 2 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0 | 0
Drooling (Nervous system disorders) | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 42 | 22 | 10 | 20
Neutropenia (Blood and lymphatic system disorders) | 5 | 4 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 22 | 11 | 6 | 12
Depression (Psychiatric disorders) | 12 | 8 | 4 | 10
Anxiety (Psychiatric disorders) | 6 | 2 | 2 | 3
Depressed mood (Psychiatric disorders) | 4 | 2 | 0 | 0
Mood swings (Psychiatric disorders) | 2 | 2 | 0 | 1
Affect lability (Psychiatric disorders) | 2 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 2
Anger (Psychiatric disorders) | 1 | 2 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 2
Apathy (Psychiatric disorders) | 1 | 1 | 0 | 0
Drug dependence (Psychiatric disorders) | 1 | 1 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Loss of libido (Psychiatric disorders) | 1 | 0 | 0 | 0
Personality disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11 | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 0 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 2 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 0 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 0
Ear infection (Infections and infestations) | 1 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 21 | 6 | 4 | 10
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 8 | 2 | 3 | 2
Photophobia (Eye disorders) | 6 | 3 | 0 | 0
Dry eye (Eye disorders) | 4 | 0 | 0 | 4
Eye pruritus (Eye disorders) | 3 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 2
Visual impairment (Eye disorders) | 0 | 2 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 1 | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 8 | 2 | 2 | 4
Lymphocyte count decreased (Investigations) | 3 | 1 | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 3
Blood pressure increased (Investigations) | 1 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 1 | 0
Blood urine present (Investigations) | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 0 | 4
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 0 | 2
Ear pruritus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Pallor (Vascular disorders) | 2 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0
Vascular pain (Vascular disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 1 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 3
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 4 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Periportal oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early at the primary efficacy endpoint (SVR12), by the sponsor on 13 January 2014 due to a decision to modify the drug development plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.